CLINICAL TRIAL: NCT06728904
Title: Intervention Effects of High-intensity Tai Chi in Mild or Moderate Asthma: a Preliminary Feasibility and Randomized Controlled Study
Brief Title: Intervention Effects of High-intensity Tai Chi in Mild or Moderate Asthma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yufen Wu, MD (Other)
Responsible Party: Sponsor-Investigator, Yufen Wu, MD, physician-in-charge, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: wuyufen2007
Record Dates: First submitted 2024-11-11; First posted 2024-12-11 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): The experimental group needs to complete high-intensity Tai Chi intervention for about 4-8 weeks according to the intervention requirements, 3-5 times/week, 45-90 minutes/time. Except for this, participants are required to participate in theoretical knowledge learning such as health lectures and online courses, as well as home autonomy exercises. This study will monitor the training status of participants through enterprise WeChat, mini programs, or app check-in to ensure high compliance. In addition, as the research subjects belong to a special population, this study expects to use the Subjective Fatigue Scale (RPE) to monitor the fatigue level of the subjects in real time to ensure safety.
  Interventions: Behavioral: Tai Chi intervention
- control group (No Intervention): This study provides health education and stretching courses for the control group. Various health education professionals will provide educational courses on asthma treatment topics, covering self-assessment, coping strategies, solutions, dietary nutrition, and disease management. At the same time, the participants in this group are required to participate in stretching courses (such as 40 minutes/time, 3 times/week), as well as home self stretching (expected to be 20 minutes/day).

INTERVENTIONS:
Behavioral: Tai Chi intervention — 40-90 minutes per session, 3-5 sessions per week. 6. Each practice mainly includes basic theoretical knowledge, warm-up exercises, standing exercises, Chen style Tai Chi, and relaxation techniques. This study expects to divide the Tai Chi intervention program into three stages: the first stage is the introductory learning of simple high-intensity Chen style Tai Chi, the second stage is the combination of strength training and Chen style Tai Chi courses, and the third stage uses optional high-intensity competitive Chen style Tai Chi or Tai Chi Sword as advanced content to consolidate learning outcomes, such as the 32 style Tai Chi Sword (HR of about 120 times/minute). The intervention plan will be combined with high-intensity interval training (HIIT) to adapt Chen style Tai Chi.
  Arms: intervention group

SUMMARY:
1、 Research objective

The main objective of this study is to investigate the therapeutic effect of a comprehensive lifestyle adjustment and stress management plan based on high-intensity Tai Chi on asthma patients. The main research areas are as follows:

1) Differences in therapeutic efficacy for mild or moderate asthma patients 2) Potential therapeutic efficacy for adult populations with different weight conditions.

2、 Research significance 2.1 Theoretical significance At present, there is limited research on the rehabilitation efficacy of high-intensity Tai Chi intervention combined with stress management programs for asthma patients. Studying the intervention effects on asthma patients among Chinese university students can fill the gap in this field and lay a theoretical foundation for further applied research in China; Exploring the application effect of high-intensity Tai Chi intervention combined with stress management plan in the treatment of asthma patients may have an important impact on improving their quality of life and rehabilitation treatment, and help expand chronic disease management strategies, which has certain theoretical value.

2.2 Practical significance The intervention effect of Tai Chi and other exercise intervention methods in the rehabilitation treatment of chronic diseases has been clinically validated and has certain innovation. This study combines this type of exercise intervention with a stress management plan, which can provide more clinical evidence and facilitate scholars to conduct other applied research, further improving the exercise rehabilitation program for asthma patients. The intervention results of exercise intervention and stress management plan for college students with asthma still have certain guiding significance for the development of rehabilitation management for asthma patients.

DETAILED DESCRIPTION:
3、 Research Methods 3.1 Main research ideas The preliminary research mainly adopts the method of literature review, completing a review of the research status, experimental methods, and measurement methods, and forming relevant theoretical foundations; The main purpose of the initial study is feasibility exploration, with a focus on evaluating participant attendance, compliance, satisfaction, and feedback. The mid-term study expanded the scope of participants and conducted a randomized controlled experiment. The study was divided into an experimental group and a control group. The experimental group received exercise intervention mainly based on Chen style Tai Chi, combined with stress management plans and health education courses. The control group received health education courses and participated in general stretching activities. Conduct data statistics for later research and propose research conclusions and recommendations based on experimental data reports.

3.2 Study Subject Selection This study focuses on asthma students from Shanghai University of Finance and Economics (including undergraduate, graduate, and doctoral students) as the subjects, and is conducted in an experimental manner. The sample size was calculated using G * power3.1 software to ensure sufficient statistical strength for this study, and the results showed that at least 20-50 subject patients need to be included.

Inclusion criteria: 1) Over 18 years old; 2) Diagnosis of mild to moderate asthma for at least 6 months (meeting the lung capacity measurement criteria for mild to moderate asthma); 3) The dosage of asthma medication has been stable for the past month (if no asthma medication has been used, it also meets the inclusion criteria).

Exclusion criteria: 1) Other lung diseases; 2) Only experiencing exercise-induced asthma (asthma is only triggered by exercise and there are no asthma symptoms in other situations; 3) pregnancy; (4) Due to chronic illness requiring oral hormone therapy in the past month; (5) Physical condition prohibits any exercise; And (6) recently unstable medical conditions. All ethnic groups and genders are eligible to participate in this study.

3.3 Main research methods 3.3.1 Experimental Method The research is generally divided into a feasibility study in the first stage and a randomized controlled study in the second stage.

The first stage feasibility study does not group the subjects, with the main purpose of testing their attendance, compliance, satisfaction, and feedback.

In the second stage of this study, participants will be randomly divided into a control group and an experimental group, and the specific tasks to be performed by both groups are as follows.

1. Research location: The study was conducted at Shanghai University of Finance and Economics;
2. Research subjects: The subjects of the feasibility study in the first stage of this research are all current students at Shanghai University of Finance and Economics, including undergraduate, graduate, and doctoral students. The second stage randomized controlled study had a wider range of participants, including not only students but also employees, teachers, and community members.
3. Testing and evaluation indicators:

   1. Feasibility indicators: Recruitment and retention: Evaluating the ability to recruit and retain participants, typically with specific goals or benchmarks (such as a retention rate of at least 70%).

      1. The proportion of all recruited personnel who persisted until the end of the intervention
      2. Attendance rate of participants during the intervention (evaluation during the intervention)
      3. The completion rate of participants' homework (evaluation during intervention)
      4. Acceptability: Evaluate the acceptability of interventions and research procedures for participants and implementers (questionnaire survey after intervention)
      5. Requirement level: Follow up evaluation after intervention to assess the extent to which new projects or interventions may be used (follow-up survey after six months of intervention)
   2. Preliminary effectiveness testing: divided into four parts: anthropometric indicators, physical health indicators, living condition indicators, and lung function indicators.

      1. Anthropometry - height, weight, waist to hip ratio, etc;
      2. Physical health indicators - grip strength, forward bending while sitting, standing on one foot, and frequency of use of emergency inhalers (average number of inhalations per day), etc;
      3. Lifestyle indicators - asthma related quality of life (through Mini Asthma Quality of Life Questionnaire, etc.) and Mood State Scale (POMS), depression and anxiety level test questionnaires, etc. These tests will be conducted before the intervention, during the second, fourth, sixth, and eighth weeks of the intervention process, and after the intervention (randomly evaluated by investigators every month for the following three months);
      4. Pulmonary function indicators - asthma control test (ACT) questionnaire, lung ventilation volume (FEV1 and PEF), and airway inflammation indicators.
4. Experimental group: The experimental group needs to complete high-intensity Tai Chi intervention for about 4-8 weeks according to the intervention requirements, 3-5 times/week, 45-90 minutes/time. Except for this, participants are required to participate in theoretical knowledge learning such as health lectures and online courses, as well as home autonomy exercises. This study will monitor the training status of participants through enterprise WeChat, mini programs, or app check-in to ensure high compliance. In addition, as the research subjects belong to a special population, this study expects to use the Subjective Fatigue Scale (RPE) to monitor the fatigue level of the subjects in real time to ensure safety.
5. Control group: This study provides health education and stretching courses for the control group. Various health education professionals will provide educational courses on asthma treatment topics, covering self-assessment, coping strategies, solutions, dietary nutrition, and disease management. At the same time, the participants in this group are required to participate in stretching courses (such as 40 minutes/time, 3 times/week), as well as home self stretching (expected to be 20 minutes/day).
6. High intensity Tai Chi intervention plan: 40-90 minutes per session, 3-5 sessions per week. 6. Each practice mainly includes basic theoretical knowledge, warm-up exercises, standing exercises, Chen style Tai Chi, and relaxation techniques. This study expects to divide the Tai Chi intervention program into three stages: the first stage is the introductory learning of simple high-intensity Chen style Tai Chi, the second stage is the combination of strength training and Chen style Tai Chi courses, and the third stage uses optional high-intensity competitive Chen style Tai Chi or Tai Chi Sword as advanced content to consolidate learning outcomes, such as the 32 style Tai Chi Sword (HR of about 120 times/minute). The intervention plan will be combined with high-intensity interval training (HIIT) to adapt Chen style Tai Chi.
7. Data testing: Researchers are responsible for organizing the testing, which is conducted by professionals. Participants conduct the experiment according to a predetermined plan.
8. Material management: The staff will prepare the corresponding experimental materials according to the experimental requirements before the start of the experiment, distribute the experimental materials to the subjects at the reception desk of the school, and archive them uniformly after the experiment to ensure that all materials have been collected. Researchers and experimenters arrive at the experimental site one hour before the start of the experiment, set up the site, and debug the experimental instruments. After the experiment, the researchers copied the test data and handed it over to the research team for backup and safekeeping.
9. Subject rewards: Participants will receive corresponding gifts as participation rewards after completing all experiments. If the subject withdraws before the completion of the experiment, the experimenter will decide whether to issue a reward based on the specific reason. The rewards will be distributed uniformly after the experiment ends.

3.3.2 Mathematical and Statistical Methods

The entered spreadsheet data was analyzed using data analysis software (SPSS 26.0, EXCEL2021, and Prism 9.0), and the main analysis methods used were:

1. Descriptive statistics: used to summarize and describe the basic information of the subjects (such as age, gender, etc.), attendance rate, intervention compliance, etc. Including mean, standard deviation, frequency distribution, etc;
2. T-test: used to compare the difference between the means of two groups, such as comparing changes in physical indicators before and after intervention;
3. Analysis of Variance (ANOVA): used to compare the mean differences between multiple groups (such as different exercise intervention intensities);
4. Multiple regression analysis: to explore the correlation between intervention effectiveness and weight, physical health, and physiological function indicators;
5. Factor analysis: to explore the impact of interventions on psychological and behavioral variables.

4、 Expected results 4.1 Chen's Tai Chi intervention combined with stress management plan intervention has a significant difference in the treatment effect on asthma patients.

4.2 There are certain differences in intervention effects among asthma patients with different body weights, physical health, and physiological function indicators.

4.3 There is a correlation between the therapeutic effect of Chen's Tai Chi intervention combined with stress management plan intervention on asthma patients and psychological and behavioral variables

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old;
2. Diagnosis of mild to moderate asthma for at least 6 months (meeting the lung capacity measurement criteria for mild to moderate asthma);
3. The dosage of asthma medication has been stable for the past month (if no asthma medication has been used, it also meets the inclusion criteria).

Exclusion Criteria:

1. Other lung diseases;
2. Only experiencing exercise-induced asthma (asthma is only triggered by exercise and there are no asthma symptoms in other situations;
3. pregnancy;
4. Due to chronic illness requiring oral hormone therapy in the past month;
5. Physical condition prohibits any exercise;
6. recently unstable medical conditions.

All ethnic groups and genders are eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1), the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration | Interventions lasting 12 weeks
  An FEV1 of less than 1 Liter indicates significant lung disease.
Peak Expiratory Flow (PEF): a person's maximum speed of expiration, measuring the airflow through the bronchi (measured in units of liters per minute) | Interventions lasting 12 weeks
  A normal peak flow in adults may be between 400 and 700 L/m. In children, a normal peak flow may range from around 150 to 450 L/m.
Asthma Control Questionnaire 7 (ACQ-7) score | Interventions lasting 12 weeks
  key measure for asthma control, assessing the adequacy of asthma control and track changes in control over time, either due to natural fluctuations or treatment interventions. It consists of seven questions that cover various aspects of asthma symptoms and their impact on daily life. To calculate the ACQ score, sum the points from all questions (1-7) and divide by 7. If question 7 is not available, sum by 6.
Perceived Stress: measured by the simplified Chinese version of the 10-item Perceived Stress Scale (SCPSS-10) | Interventions lasting 12 weeks
  The Simplified Chinese version of the 10-item Perceived Stress Scale (SCPSS-10) has been used to measure and evaluate perceived stress in various populations. This scale allows researchers to assess stress levels effectively among Chinese-speaking individuals. See Huang, F. et al, 2020. Psychometric properties of the perceived stress scale in a community sample of Chinese. BMC psychiatry, 20, pp.1-7.
Feasibility (measured by attendance rate of the training sessions) | Measured throughout the 12 weeks of intervention
  Feasibility in terms of attendance rate for training sessions is often assessed by setting a benchmark, such as achieving over 50% attendance. Higher attendance rates generally indicate greater feasibility and engagement with the training program. Low attendance can suggest issues with the program's design or relevance, especially in unsupervised training interventions, which tend to have lower attendance and effectiveness.

SECONDARY OUTCOMES:
Grip strength by kilograms | Interventions lasting 12 weeks
  Measured by a grip strength tester (for individuals aged 10-80), the average grip strength is approximately 37.2 kg for the right hand and 34.7 kg for the left hand.

CONTACTS AND LOCATIONS:
Overall Officials: Yufen Wu, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai University of Finance and Economics, Shanghai, China

IPD SHARING:
Plan to Share IPD: No